CLINICAL TRIAL: NCT04283526
Title: A Phase Ib, Multicenter, Open-label Dose Escalation and Expansion Platform Study of Select Combinations in Adult Patients With Myelofibrosis
Brief Title: Study of Select Combinations in Adults With Myelofibrosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was cancelled before enrolling any patients for business related reasons.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CMBG453D12101; 2019-003738-18 (EudraCT Number)
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Primary Myelofibrosis; Myelofibrosis; PMF; Post-Essential Thrombocythemia Myelofibrosis; Post-Polycythemia Vera Myelofibrosis
Keywords: Post-essential thrombocythemia myelofibrosis; PET-MF; MF; myeloproliferative neoplasms; thrombocythemia myelofibrosis; polycythemia vera; essential thrombocythemia; primary myelofibrosis; Myelofibrosis (PMF); Post-Polycythemia Vera Myelofibrosis (PPV-MF); Post-Essential Thrombocythemia Myelofibrosis (PET-MF); primary myelofibrosis (PMF); osteomyelofibrosis; myeloproliferative neoplasm; chronic idiopathic myelofibrosis (cIMF); Angnogenic myeloid metaplasia; myelofibrosis with myeloid metaplasia (MMM)
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders; Polycythemia Vera; Thrombocythemia, Essential | interventions — sabatolimab; NIS-793; spartalizumab; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- NIS793 + MBG453 (Experimental): treatment with NIS793 + MBG453
  Interventions: Drug: MBG453; Drug: NIS793
- NIS793 + MBG453 + Spartalizumab (Experimental): Treatment with NIS793 + MBG453 + Spartalizumab
  Interventions: Drug: MBG453; Drug: NIS793; Drug: Spartalizumab
- NIS793 + MBG453 + Decitabine (Experimental): treatment with NIS793 + MBG453 + Decitabine
  Interventions: Drug: MBG453; Drug: NIS793; Drug: Decitabine
- NIS793 (Experimental): treatment with NIS793
  Interventions: Drug: NIS793
- MBG453 (Experimental): treatment with MBG453
  Interventions: Drug: MBG453

INTERVENTIONS:
Drug: MBG453 — Intravenous. 600mg. Every first day of a 21-day cycle, or on days 8 and 29 of a 42-day cycle (when in combination with Decitabine).
  Arms: MBG453; NIS793 + MBG453; NIS793 + MBG453 + Decitabine; NIS793 + MBG453 + Spartalizumab
Drug: NIS793 — Intravenous. 2100mg. Every first day of a 21-day cycle, or on days 8 and 29 of a 42-day cycle (when in combination with Decitabine).
  Arms: NIS793; NIS793 + MBG453; NIS793 + MBG453 + Decitabine; NIS793 + MBG453 + Spartalizumab
Drug: Spartalizumab — Intravenous. 300mg. Every first day of a 21-day cycle
  Other Names: PDR001
  Arms: NIS793 + MBG453 + Spartalizumab
Drug: Decitabine — Intravenous. Starting dose: 5mg/m2 (dose cap at 20mg/m2). On days 1, 2 and 3 of a 42-day cycle
  Other Names: Dacogen
  Arms: NIS793 + MBG453 + Decitabine

SUMMARY:
The purpose of this study is to investigate the safety, pharmacokinetics (PK) and preliminary efficacy of both the combination of MBG453 and NIS793 with or without decitabine or spartalizumab as well as single agent MBG453 and/or NIS793 single agent in myelofibrosis (MF) subjects post treatment with a Janus Kinase (JAK) inhibitor.

In this study, combination therapies with novel agents including immune therapy will focus on determining the promising combinations that provide acceptable safety and efficacy independent of JAK inhibitors. Immune therapy combinations, such as MBG453 in combination with NIS793, might offer the potential to target MF across genetic heterogeneity.

The primary objective of this study is to characterize the safety, tolerability and recomended dose for each treatment combination (MBG453 + NIS793, MBG453 + NIS793 + decitabine, and MBG453 + NIS793 + spartalizumab)

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety, pharmacokinetics (PK) and preliminary efficacy of both the combination of MBG453 and NIS793 with or without decitabine or spartalizumab as well as single agent MBG453 and/or NIS793 single agent in myelofibrosis (MF) subjects post treatment with a Janus Kinase (JAK) inhibitor.

In this study, combination therapies with novel agents including immune therapy will focus on determining the promising combinations that provide acceptable safety and efficacy independent of JAK inhibitors. Immune therapy combinations, such as MBG453 in combination with NIS793, might offer the potential to target MF across genetic heterogeneity.

The primary objective of this study is to characterize the safety, tolerability and recomended dose for each treatment combination (MBG453 + NIS793, MBG453 + NIS793 + decitabine, MBG453 + NIS793 + spartalizumab).

Secondary Objectives are: to evaluate the efficacy based on the revised International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) response criteria, to evaluate the effect of each combination treatment in delaying progression of MF and estimate time to progression free survival (PFS) event, and to characterize the PK profile of each treatment arm Study is designed as a Phase Ib, multi center, open label study with multiple treatment arms. The study is comprised of a dose evaluation/escalation part and a dose expansion part.

MBG453 in combination with NIS793 will be explored as the initial backbone. As the study progresses and based on emerging clinical data collected from this study, Novartis, in agreement with the study Investigators will decide whether or not:

* To proceed with any treatment arm that reaches recommended dose(s) to explore further the safety, tolerability, and anti-tumor activity in the dose expansion part.
* To add a third partner to comprise a triplet treatment arm in the dose evaluation/escalation part (such as Treatment Arm 2 with decitabine or Treatment Arm 3 with spartalizumab.
* To explore MBG453 single agent (Treatment Arm 4) and/or NIS793 single agent (Treatment Arm 5) in the dose expansion part in order to assess the single agent contributions to efficacy.

The patient population will include male or female adults (age 18 or over) with a confirmed diagnosis of primary myelofibrosis (PMF) as defined by the World Health Organization (WHO) criteria, or Post-Polycythemia Vera Myelofibrosis (PPV-MF), or Post-Essential Thrombocythemia Myelofibrosis (PET-MF) based on the revised IWG-MRT) criteria, irrespective of JAK2 mutation status and must have been treated with a JAK inhibitor for at least 28 days but no more than 6 months and experienced according to the Investigator suboptimal response defined by loss of spleen response, or worsening of symptoms or discontinuation due to adverse events (AE).

Data analysis: the primary objective of the study is to characterize the safety and tolerability of each combination and identify the recommended dose. The primary analysis will be based on a Bayesian Hierarchical Logistic Regression Model (BHLRM) and summaries of other safety, tolerabitliy endpoints. Efficacy will be assessed based on IWG-MRT. The study data will be analyzed and reported based on all patients' data up to the time when 80% of the patients have completed the follow-up for disease progression or discontinued the study for any reason, and all patients have completed treatment and the safety follow-up period.

ELIGIBILITY:
Key inclusion criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Male or female subjects must be ≥ 18 years of age at the time of signing the informed consent form (ICF).
3. Subjects have a diagnosis of PMF as defined by the WHO criteria, or diagnosis of PET-MF or PPV-MF as defined by the IWG-MRT criteria (International Working Group for Myelofibrosis Research and Treatment).
4. Subjects must have been treated with a JAK inhibitor for ≥3 months with inadequate efficacy response defined as <10% spleen volume reduction by MRI or <30% decrease from baseline in spleen length by physical examination or regrowth to these parameters following an initial response.

   And/or

   Treatment for ≥28 days complicated by either:
   * Development of a red blood cell transfusion requirement (at least 2 units/month for 2 months); or
   * Grade ≥3 AEs of thrombocytopenia, anemia, hematoma, and/or hemorrhage while on treatment with JAK inhibitor.
5. Palpable spleen of at least 5 cm from the LCM to the point of greatest splenic protrusion or enlarged spleen volume of at least 450 cm3 per MRI or CT scan at baseline (an MRI/CT scan up to 8 weeks prior to first dose of study treatment can be accepted).
6. Absolute neutrophil count (ANC) ≥ 1000/μL.
7. Dose evaluation / Dose escalataion: Platelet count ≥ 75,000/μL without transfusion support Dose expansion: Platelet count ≥ 50,000/μL without transfusion support.

Key exclusion criteria:

1. Subjects with Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS), or peripheral blasts ≥ 10 %, or AML transfromed from previous MPN.
2. Subjects having received JAK inhibitors, systemic antineoplastic therapy (including unconjugated therapeutic antibodies, toxin immunoconjugates, and alpha-interferon) or any experimental therapy within 14 days or five half-lives, whichever is shorter, before the first dose of study treatment.
3. Prior autologous or allogeneic stem cell transplant at any time.
4. Candidate for allogenic hematopoietic stem cell transplantation at the time of enrolment.
5. Splenic irradiation within 6 months prior to the first dose of study treatment.
6. Prior splenectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2024-04-11 (Estimated); Study Completion 2024-04-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose limiting toxicities (DLT) | 12 months
  A dose-limiting toxicity (DLT) is defined as a clinically relevant adverse event or abnormal laboratory value where the relationship to study treatment cannot be ruled out, and which is unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the DLT monitoring period and meets any of the criteria included in Table 6-4 (Criteria for defining dose-limiting toxicities).
Incidence and severity of AEs and SAEs, including changes in laboratory values, vital signs, and ECGs | 36 months
  Incidence and severity of AEs and SAEs, including changes in laboratory values, vital signs, and electrocardiograms (ECGs). A Serious adverse event (SAE) is defined as one of the following:
  * Is fatal or life-threatening
  * Results in persistent or significant disability/incapacity
  * Constitutes a congenital anomaly/birth defect
  * Is medically significant
  * Requires inpatient hospitalization or prolongation of existing hospitalization.
Dose interruptions | 36 months
  Tolerability measured by the number of subjects who have interruptions of study treatment and reason for interruptions
Dose reductions | 36 months
  Tolerability measured by the number of subjects who have reductions of study treatment and reason for reductions
Dose intensity | 36 montths
  Tolerability measured by the dose intensity of study drug, Relative Dose intensity for subjects with non-zero duration of exposure is computed as the ratio of dose intensity and planned dose intentity

SECONDARY OUTCOMES:
Clinical benefit rate based on revised IWG-MRT (International Working Group Myelofibrosis Research & Treatment) criteria: complete response (CR), partial response (PR), stable disease, progressive disease (PD), Anemia response, Spleen response, relapse | 36 months
  Proportion of subjects achieving IWG-MRT (International Working Group for Myelofibrosis Research and Treatment) response criteria:
  * Proportion of subjects with: complete response (CR) and partial response (PR), stable disease, progressive disease (PD).
  * Proportion of subjects achieving Anemia response (anemia improvement of Hb ≥2.0 g/dL for transfusion independent subjects at baseline; or transfusion independence for transfusion dependent subjects at baseline).
  * Proportion of subjects achieving spleen response (by palpation) from baseline or spleen volume reduction (by imaging) from baseline.
  * Proportion of subjects experiencing relapse.
Proportion of subjects achieving improvement of Anemia | 36 months
  Proportion of subjects achieving improvement of Hb level of ≥ 1.5 g/dL from baseline
Progression-free survial time (PFS) | 36 months
  PFS is defined as the time from the date of start of treatment to the date of death by any cause or date of first documented progression as per IWG-MRT (International Working Group for Myelofibrosis Research and Treatment) criteria:
  * Progressive splenomegaly as assessed by increasing spleen volume (by MRI/CT) of ≥ 25% from baseline.
  * Accelerated phase defined by a circulating peripheral blood blast content of > 10% but <20% confirmed after 2 weeks.
  * Deteriorating cytopenia (dCP) independent from treatment, defined for all patients by platelet count < 35 x10^9/L or neutrophil count < 0.75 x10^9/L that lasts for at least 4 weeks.
  * Leukemic transformation defined by a peripheral blood blast content of ≥ 20% associated with an absolute blast count of ≥ 1x10^9/L that lasts for at least 2 weeks or a bone marrow blast count of ≥ 20%.
Duration of response | 36 months
  Time between the date of first documented response (as per the revised International Working Group for Myelofibrosis Research and Treatment IWG-MRT criteria) and the date of first documented progression or death.
Cmax (Maximum Concentration) | 36 months
  The maximum observed plasma, blood serum or other body fluid drug concentration
Tmax | 36 months
  Time to reach maximum plasma, blood serum or other body fluid drug concentration

CONTACTS AND LOCATIONS:
Overall Officials: Alesandro Pastore Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No